CLINICAL TRIAL: NCT02929095
Title: The Effect of Remifentanil-dexmedetomidine Compared With Remifentanil-midazolam on Patient's Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2016-0701
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Dexmedetomidine; Midazolam; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients in the dexmedetomidine group (Experimental): Patients in the dexmedetomidine group are given 1 μg/kg/h of dexmedetomidine for 10 minutes on initiation of the procedure and then 0.2-0.7 μg/kg/h until end of the procedure and are given 1.2-7.2 μg/kg/h of remifentanil until end of the procedure
  Interventions: Drug: dexmedetomidine; Drug: remifentanil
- Patients in the midazolam group (Active Comparator): Patients in the midazolam group are given midazolam 0.02-0.05mg/kg bolus on initiation of the procedure and are given 1.2-7.2 μg/kg/h of remifentanil until end of the procedure
  Interventions: Drug: midazolam; Drug: remifentanil

INTERVENTIONS:
Drug: dexmedetomidine
  Arms: Patients in the dexmedetomidine group
Drug: midazolam
  Arms: Patients in the midazolam group
Drug: remifentanil — - remifentanil will be administered to both dexmedetomidine and midazolam group as a routine part of procedure and it is no of interest of the protocol

SUMMARY:
Percutaneous trans-arterial angioplasty(PTA) is one of the peripheral arterial occlusive disease(PAOD) treatment. During and after PTA, ischemia-reperfusion pain is induced so proper analgesia is important. ischemia-reperfusion injury is due to reactive oxygen species. Dexmedetomidine has analgesic, sedative and anti oxidant effect. So the investigators research the patient's satisfaction that are given the dexmedetomidine during PTA procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo percutaneous trans-arterial angioplasty
* American Society of Anesthesiologists (ASA) class I, II, III

Exclusion Criteria: Subjects are ineligible if they have the below condition

* psychiatric medication
* myocardial infarction within 1 year
* cardiac surgery within 1 year
* heart failure
* fever (>38 degree)
* uncontrolled hypertension
* cognitive dysfunction
* disabling mental change disorder
* being unable to communicate or speak Korean

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
patient's satisfaction | 1 hour after the procedure (PTA)
  patient's satisfaction is measured by 5-point numerical rating scale ((0=extremely dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, and 4=extremely satisfied)
patient's satisfaction | 6 hours after the procedure (PTA)
  patient's satisfaction is measured by 5-point numerical rating scale ((0=extremely dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, and 4=extremely satisfied)
patient's satisfaction | 12 hours after the procedure (PTA)
  patient's satisfaction is measured by 5-point numerical rating scale ((0=extremely dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, and 4=extremely satisfied)
patient's satisfaction | 24 hours after the procedure (PTA)
  patient's satisfaction is measured by 5-point numerical rating scale ((0=extremely dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, and 4=extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea